CLINICAL TRIAL: NCT01453634
Title: A Randomized, Open Label, Four Week, Pharmacodynamic/Pharmacokinetic, Efficacy, and Safety Study of Lunacalcipol (CTA018) Injection in Subjects With Stage 5 Chronic Kidney Disease With Secondary Hyperparathyroidism on Hemodialysis
Brief Title: Four Week, Pharmacodynamic/Pharmacokinetic, Efficacy, and Safety Study of Lunacalcipol (CTA018)
Acronym: 2007
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The company is no longer pursuing this study.
Sponsor: OPKO Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTA018-2007
Record Dates: First submitted 2011-10-13; First posted 2011-10-18 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2014-09

CONDITIONS: Stage 5 Chronic Kidney Disease (CKD); Secondary Hyperparathyroidism (SHPT); Hemodialysis (HD)
Keywords: chronic kidney disease (CKD); secondary hyperparathyroidism (SHPT); hemodialysis (HD)
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperparathyroidism, Secondary

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lunacalcipol 180 (Experimental): 180 µg (n=4)Lunacalcipol Injection
  Interventions: Drug: Lunacalcipol 180
- Lunacalcipol 270 (Experimental): 270 µg (n=8)Lunacalcipol Injection
  Interventions: Drug: Lunicalcipol 270

INTERVENTIONS:
Drug: Lunacalcipol 180 — 4 subjects are planned to receive a total of 11 doses of the study drug given three times per week (tiw) over 24 days (day 1 to day 24), administered not more often than every other day.
  Arms: Lunacalcipol 180
Drug: Lunicalcipol 270 — 8 subjects are planned to receive a total of 11 doses of the study drug given three times per week (tiw) over 24 days (day 1 to day 24), administered not more often than every other day.
  Arms: Lunacalcipol 270

SUMMARY:
Open-label, pharmacodynamic, safety, pharmacokinetic and efficacy study of Lunacalcipol Injection.

DETAILED DESCRIPTION:
This is a prospective, open-label, PD, safety, PK and efficacy study of Lunacalcipol Injection. Approximately 12 subjects will be randomized into 1 of 2 treatment groups receiving either 180 µg (n=4) or 270 µg (n=8) Lunacalcipol Injection in a 1:2 ratio, respectively. All subjects are planned to receive a total of 11 doses of the study drug given three times per week (tiw) over 24 days (day 1 to day 24), administered not more often than every other day.

Previously defined criteria relating to serum levels of iPTH, Ca, and P will be reviewed by the Medical Monitor to determine subject safety. If any of the criteria are observed, subjects will be discontinued from the study, receiving no further administration of the study drug and will be followed for safety. Safety data will be reviewed by the Medical Monitor for the first 2 subjects in the 270 µg group. If the first 2 subjects meet dose group discontinuation criteria, including treatment emergent calciphylaxis, treatment-emergent adverse events (TEAEs) related to elevated serum Ca levels, or a reported death associated with elevated serum Ca levels or related to study drug, subjects beyond the first 2 will not be dosed.

A Data and Safety Monitoring Board (DSMB) will be appointed to provide an independent evaluation of all safety data, including all laboratory results and serious adverse events (SAEs). The DSMB will conduct its review after 4 subjects in the 270 µg dose group have completed at least 6 doses, at any time death is reported, or at the request of the DSMB. The DSMB will also conduct an additional review at the End of Study.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have a body mass index (BMI) between 18 and 35 kg/m2, inclusive.
* Prior to study entry, subjects must be undergoing maintenance HD tiw, be in stable condition (ie, on maintenance HD for at least 8 weeks) and be expected to remain on HD for the duration of the study.
* Subject must be willing and able to discontinue vitamin D and/or bone metabolism therapy for a minimum 2 week wash-out prior to administration of study drug and through the EOS visit. This includes vitamin D supplements daily dose containing more than 1000 IU of ergocalciferol or cholecalciferol) and analogs (calcitriol, paricalcitol, doxercalciferol), cinacalcet, teriparatide, calcitonin, maintenance glucocorticoids (greater than a prednisone equivalent of 5 mg/day), selective estrogen receptor modulators (SERMs; raloxifene or tamoxifen) or other drugs that may affect Ca metabolism.
* Subjects must not have taken bisphosphonates for at least 3 months (90 days) prior to the first dose of study drug.
* Subject laboratory values must be within the following ranges:

  * Plasma iPTH ≥350 pg/mL (35 pmol/L) and <1000 pg/mL (100 pmol/L)
  * Total serum Ca ≥8.4 mg/dL (2.1 mmol/L) and <10.0 mg/dL (2.5 mmol/L)
  * Serum P ≥2.5 mg/dL (0.8 mmol/L) and <6.2 mg/dL (2.0 mmol/L)
* Total serum 25-hydroxyvitamin D level at screening must be ≥15 ng/mL (37 nmol/L).
* Subject must be willing and able to comply with study instructions and commit to all clinic visits for the duration of the study.
* Female subjects of childbearing potential must be neither pregnant nor lactating and must have a negative serum pregnancy test at screening and agree to use effective contraception (implants, injectables, combined oral contraceptives, intrauterine device (IUD), sexual abstinence, or vasectomized partner) for the duration of the study.

Exclusion Criteria:

* Subject cannot have clinically significant liver disease (alanine aminotransferase [ALT], aspartate amino transferase [AST] or bilirubin > 2x ULN), or any clinical evidence of significant hepatic dysfunction during the screening period deemed clinically significant by the investigator.
* Subject cannot be currently taking cytochrome P450 3A inhibitors (eg, ketoconazole or erythromycin) or P450 3A inducers.
* Subject cannot have a known history of kidney stones within the previous 2 years.
* Subject cannot have a known previous or concomitant serious illness or medical condition, such as malignancy, human immunodeficiency virus (HIV) or hepatitis that in the opinion of the investigator may worsen and/or interfere with participation in the study.
* Subject cannot have a history of neurological/psychiatric disorders, including psychotic disorders or dementia, or any other reason, which in the opinion of the investigator makes adherence to a regular treatment or follow-up schedule unlikely.
* Subject cannot have any clinically significant abnormalities, as determined by the investigator, based on a 12-lead ECG, PE and laboratory assessments conducted during screening.
* Subject cannot have a known or suspected hypersensitivity to any of the constituents of the investigational product.
* Subject cannot be currently participating in or have participated in an interventional/investigational study within 30 days prior to the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-01; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Measure the intact parathyroid hormone (iPTH) levels following Lunacalcipol Injection | 3 screening visits will occur within up to 42 days, Subjects will receive a total of 11 doses of study drug given 3 times weekly over 24 days. Following 24 days of treatment, subjects will undergo 2 days of follow-up and an end of study (EOS) assessment.

SECONDARY OUTCOMES:
Assess the safety of Lunacalcipol Injection | 3 screening visits will occur within up to 42 days, Subjects will receive a total of 11 doses of study drug given 3 times weekly over 24 days. Following 24 days of treatment, subjects will undergo 2 days of follow-up and an end of study (EOS) assessment.
  Criteria relating to serum levels of iPTH, Ca, and P will be reviewed by the Medical Monitor. If any of the criteria are observed, subjects will be discontinued from the study and will be followed for safety. Safety data will be reviewed by the Medical Monitor for the first 2 subjects in the 270 µg group. If the first 2 subjects meet dose group discontinuation criteria, subjects beyond the first 2 will not be dosed.